CLINICAL TRIAL: NCT04663594
Title: An Online Cultural Experience to Support Mental Health in People Aged 16-24 During COVID-19: the O-ACEPOP (Online Active Community Engagement Proof of Principle) Study
Brief Title: Online Culture for Mental Health in People Aged 16-24
Acronym: O-ACEPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0009275
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two arm study, 1:1 randomisation (stratified by gender)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ways of Being online Experience (Experimental): Ways of Being (WoB) every day for three days
  Interventions: Other: WofB
- Ashmolean Website (Other): The Ashmolean Website every day for three days
  Interventions: Other: Ashmolean Website

INTERVENTIONS:
Other: WofB — Online experience designed to reduce anxiety and depression and support mental health and wellbeing
  Arms: Ways of Being online Experience
Other: Ashmolean Website — A generic museum website owned by the Ashmolean Museum of Art and Archaeology at the University of Oxford.
  Arms: Ashmolean Website

SUMMARY:
O-ACE POP is a randomised controlled trial of an online cultural experience named Ways of Being, compared to a typical museum website (the Ashmolean Museum). The primary aim is to compare these two interventions by efficacy on mood, distress (depression and anxiety), flourishing and investigate potential mechanisms of action, as well as the feasibility of a larger scale RCT.

DETAILED DESCRIPTION:
People of target age will be actively recruited with a link to Participant information and E-consent procedures for those who fulfil inclusion criteria and consent to entering their email address.

Consenting participants will enter a demographic questionnaire. Participants will then be emailed a unique ID number and requested to complete a baseline assessment on a computer, including self-report measures and online tasks. Participants will then be randomised to WoB or the Ashmolean Website. Once randomised participants will be requested to log on to the intervention at least once a day for the next three days

Randomisation and blinding Randomisation procedures will be followed. The participants will be aware of which intervention they have been allocated to. All measures are online and self-report.

Ways of Being (WoB) is an online cultural experience designed to reduce distress (symptoms of anxiety and depression) and promote positive mental health in people aged 16-24. It is a web-experience based on qualitative research and co-production with people aged 16-24. The experience is based on human centred narratives related to the objects and artworks of the Ashmolean Museum in Oxford and partner museums. In addition, other people's viewpoints on the objects and artworks or narrative, are a focus of the experience. The experience combines text, audio and aesthetic elements.

The Ashmolean Website is a generic museum website owned by the Ashmolean Museum of Art and Archaeology at the University of Oxford. The Ashmolean is the oldest public museum in the UK, and has incredibly rich and diverse collections from around the globe, ranging from classical civilisation to the Pre-Raphaelites and modern art. The website is aimed at general museum visitors, tourists, families, primary, secondary and tertiary learners, teachers, and those with specialist cultural interests.

Statistical Analysis Plan The main outcome will be the mean PANAS score at each time point. These will be regressed on time (pre-intervention vs. during, exit and follow up), a group indicator (WoB vs. the Ashmolean Website), and their interaction.

ELIGIBILITY:
Inclusion Criteria:

People ages 16-24

Exclusion Criteria:

* No access to a laptop or desktop computer

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 463 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
PANAS | Baseline, Days 2-4 (morning and evening), Day 5, six weeks
  Is a widely used scale of emotion and comprises 20 items, 10 measuring positive affect (excited, inspired etc) and 10 measuring negative affect (upset, afraid etc), on a Likert Scale of 1 (very slightly) to 5 (extremely). We will be measuring change between baseline and time-points (in Timeframe)
K10 | Baseline, Day 5, six weeks
  The K10 is a well validated self-report measure of distress (depression and anxiety). We will be measuring change between baseline and time-points (in Timeframe)

SECONDARY OUTCOMES:
Facial expression recognition task | Baseline, Day 5, six weeks
  The facial expression recognition task provides an objective measure of emotional bias which is associated with vulnerability to depression. We will be measuring change between baseline and time-points (in Timeframe)
Probabilistic Incentive Learning Task | Baseline, Day 5, six weeks
  This is an instrumental learning task in which the participant gains or loses points by choosing between two paired images. The participant is told that some images are more likely (but not always) to be associated with gains and some with losses. The explicit aim is to maximize points. We will be measuring change between baseline and time-points (in Timeframe)
Flourishing | Baseline, Day 5, six weeks
  The Flourishing Scale is an 8-item measure of self-perceived success in domains such as self-esteem, relationships, optimism and purpose. We will be measuring change between baseline and time-points (in Timeframe)
Loneliness | Baseline, Day 5, six weeks
  The UCLA Loneliness Scale is a self-report inventory that uses a Likert-type scale to assess subjective feelings of loneliness. In addition we will add an item directly asking about loneliness. We will be measuring change between baseline and time-points (in Timeframe).

CONTACTS AND LOCATIONS:
Locations (1):
- Ashmolean Museum Website, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available on OSF once peer reviewed
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available on OSF once peer reviewed

REFERENCES:
- [Derived] Syed Sheriff RJ, Vuorre M, Riga E, Przybylski AK, Adams H, Harmer CJ, Geddes JR. A cultural experience to support mental health in people aged 16-24 during the COVID-19 pandemic compared to a typical museum website: study protocol of an online randomised controlled trial. Trials. 2021 Jul 22;22(1):482. doi: 10.1186/s13063-021-05441-z. PMID 34294126